CLINICAL TRIAL: NCT00553267
Title: An Eight-week Randomised, Double-blind Study to Compare the Fixed-dose Combination of Telmisartan 40mg + Amlodipine 10mg Versus Telmisartan 80mg + Amlodipine 10mg Versus Amlodipine 10mg Monotherapy in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Amlodipine 10mg Monotherapy
Brief Title: Telmisartan/Amlodipine (80/10) vs. Telmisartan/Amlodipine (40/10) vs. amlodipine10 in Resistant Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1235.6; EUDRACT 2007-002421-68
Record Dates: First submitted 2007-10-08; First posted 2007-11-05 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

INTERVENTIONS:
Drug: fixed dose combination of telmisartan+amlodipine
Drug: amlodipine

SUMMARY:
The primary objective of this trial is to demonstrate that the fixed dose combination of telmisartan 40mg + amlodipine 10mg (T40/A10) or the fixed dose combination of telmisartan 80mg + amlodipine 10mg (T80/A10) is superior in reducing blood pressure at eight weeks compared with amlodipine 10mg monotherapy (A10) in patients who fail to respond to six weeks treatment with A10.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of essential hypertension and blood pressure not adequately controlled before informed consent (inadequate control defined as seated diastolic blood pressure (DBP) >= 95 mmHg if on existing antihypertensive treatment or seated DBP >= 100 mmHg if treatment-naïve).
* failure to respond to six weeks treatment with amlodipine 10mg. (Failure to respond defined as seated DBP >= 90 mmHg.)
* able to stop any current antihypertensive therapy without unacceptable risk to the patient.
* willing and able to provide written informed consent.

Exclusion Criteria:

* pregnancy, breast-feeding, unwilling to use effective contraception (if female of child-bearing potential).
* known or suspected secondary hypertension.
* mean seated systolic blood pressure (SBP) >=200 mmHg and/or mean seated DBP >= 120 mmHg during run-in treatment or mean seated SBP >= 180 mmHg and/or mean seated DBP >= 120 mmHg at the randomisation visit or at any time during randomised treatment.
* any clinically significant hepatic impairment or severe renal impairment bilateral renal artery stenosis or renal artery stenosis in a solitary kidney or post post-renal transplant.
* clinically relevant hyperkalaemia.
* uncorrected volume or sodium depletion.
* primary aldosteronism.
* hereditary fructose or lactose intolerance.
* symptomatic congestive heart failure.
* patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or ARBs.
* history of drug or alcohol dependency within the six months prior to signing consent.
* concurrent participation in another clinical trial or any investigational therapy within thirty days prior to signing consent.
* hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve.
* known allergic hypersensitivity to any component of the formulations under investigation. (Includes known hypersensitivity to telmisartan or other ARBs or amlodipine or other dihydropyridine CCBs.)
* non-compliance with study medication (defined as less than 80% or more than 120%) during the open-label run-in treatment period.
* current treatment with any antihypertensive agents, whether or not prescribed for this indication, that cannot be safely stopped (investigator¿s decision) by the start of the run-in period.
* chronic administration of any medication known to affect blood pressure, other than the trial medication.
* any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan and amlodipine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (97):
- Australia (5):
  - 1235.6.61003 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1235.6.61004 Boehringer Ingelheim Investigational Site, Liverpool, New South Wales
  - 1235.6.61002 Boehringer Ingelheim Investigational Site, Kippa-Ring, Queensland
  - 1235.6.61001 Boehringer Ingelheim Investigational Site, Milton, Queensland
  - 1235.6.61005 Boehringer Ingelheim Investigational Site, Elizabeth Vale, South Australia
- Austria (6):
  - 1235.6.43007 Boehringer Ingelheim Investigational Site, Eggenburg
  - 1235.6.43006 Boehringer Ingelheim Investigational Site, Hainburg A.d. Donau
  - 1235.6.43005 Boehringer Ingelheim Investigational Site, Hartberg
  - 1235.6.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1235.6.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1235.6.43003 Boehringer Ingelheim Investigational Site, Vienna
- Bulgaria (10):
  - 1235.6.35912 Boehringer Ingelheim Investigational Site, Burgas
  - 1235.6.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35905 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35907 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35910 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35911 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.6.35901 Boehringer Ingelheim Investigational Site, Varna
- Czechia (7):
  - 1235.6.42002 Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - 1235.6.42006 Boehringer Ingelheim Investigational Site, Brno
  - 1235.6.42001 Boehringer Ingelheim Investigational Site, Pilsen
  - 1235.6.42003 Boehringer Ingelheim Investigational Site, Prague
  - 1235.6.42004 Boehringer Ingelheim Investigational Site, Příbram
  - 1235.6.42005 Boehringer Ingelheim Investigational Site, Slaný
  - 1235.6.42007 Boehringer Ingelheim Investigational Site, Strakonice
- Ireland (6):
  - 1235.6.35304 Wilmer Road, Birr
  - 1235.6.35305 Dr. Ger McLaughlin, Carrigtohill
  - 1235.6.35302 Slaney Medical Centre, Enniscorthy
  - 1235.6.35303 Gorey Medical Centre, Coral House,, Gorey
  - 1235.6.35306 The Red House Surgery, Mallow
  - 1235.6.35301 Boehringer Ingelheim Investigational Site, New Ross
- Italy (3):
  - 1235.6.39002 Boehringer Ingelheim Investigational Site, Broni (pv)
  - 1235.6.39006 Boehringer Ingelheim Investigational Site, Coppito (AQ)
  - 1235.6.39001 Boehringer Ingelheim Investigational Site, Ferrara
- New Zealand (3):
  - 1235.6.64003 Boehringer Ingelheim Investigational Site, Dunedin
  - 1235.6.64002 Boehringer Ingelheim Investigational Site, Otahuhu, Auckland
  - 1235.6.64001 Boehringer Ingelheim Investigational Site, Tauranga
- Russia (9):
  - 1235.6.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70007 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70009 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.6.70010 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.6.70011 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.6.70012 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (7):
  - 1235.6.42103 Boehringer Ingelheim Investigational Site, Dolný Kubín
  - 1235.6.42106 Boehringer Ingelheim Investigational Site, Kralovsky Chmlec
  - 1235.6.42104 Boehringer Ingelheim Investigational Site, Liptovský Mikuláš
  - 1235.6.42102 Boehringer Ingelheim Investigational Site, Považská Bystrica
  - 1235.6.42105 Boehringer Ingelheim Investigational Site, Prešov
  - 1235.6.42101 Boehringer Ingelheim Investigational Site, Trenčín
  - 1235.6.42107 Boehringer Ingelheim Investigational Site, Vráble
- Spain (7):
  - 1235.6.34008 Hospital Municipal de Badalona, Badalona
  - 1235.6.34009 Boehringer Ingelheim Investigational Site, Barcelona
  - 1235.6.34001 Hospital Gral de Jerez de la Frontera, Jerez de La Frontera (Cádiz)
  - 1235.6.34006 C.A.P. Mossen Cinto Verdaguer, L'Hospitalet de Llobregat (Barcelona)
  - 1235.6.34003 Hospital Doce de Octubre, Madrid
  - 1235.6.34004 Hospital La Princesa, Madrid
  - 1235.6.34011 Boehringer Ingelheim Investigational Site, Santa Coloma de Gramanet
- 1235.6.41005 Boehringer Ingelheim Investigational Site, Gordola, Switzerland
- Turkey (Türkiye) (4):
  - 1235.6.90004 Boehringer Ingelheim Investigational Site, Erzurum
  - 1235.6.90003 Boehringer Ingelheim Investigational Site, Istanbul
  - 1235.6.90005 Boehringer Ingelheim Investigational Site, Istanbul
  - 1235.6.90001 Boehringer Ingelheim Investigational Site, Izmir
- Ukraine (13):
  - 1235.6.38010 Boehringer Ingelheim Investigational Site, Dnipro
  - 1235.6.38001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.6.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.6.38008 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.6.38011 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.6.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.6.38006 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.6.38012 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.6.38013 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.6.38002 Boehringer Ingelheim Investigational Site, Lviv
  - 1235.6.38005 Boehringer Ingelheim Investigational Site, Odesa
  - 1235.6.38009 Boehringer Ingelheim Investigational Site, Odesa
  - 1235.6.38007 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (16):
  - 1235.6.44010 Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - 1235.6.44008 Boehringer Ingelheim Investigational Site, Blackpool
  - 1235.6.44016 Boehringer Ingelheim Investigational Site, Blackpool
  - 1235.6.44011 Boehringer Ingelheim Investigational Site, Burbage, Hinkley
  - 1235.6.44007 Boehringer Ingelheim Investigational Site, Chestfield, Whitstable
  - 1235.6.44005 Boehringer Ingelheim Investigational Site, Chorley
  - 1235.6.44002 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 1235.6.44009 Boehringer Ingelheim Investigational Site, Ely
  - 1235.6.44001 Boehringer Ingelheim Investigational Site, Fowey
  - 1235.6.44003 Boehringer Ingelheim Investigational Site, Glasgow
  - 1235.6.44012 Boehringer Ingelheim Investigational Site, Penzance
  - 1235.6.44013 Boehringer Ingelheim Investigational Site, Plymouth
  - 1235.6.44004 Boehringer Ingelheim Investigational Site, Reading
  - 1235.6.44015 Boehringer Ingelheim Investigational Site, Saint Stephen, Saint Austell
  - 1235.6.44014 Boehringer Ingelheim Investigational Site, Saltash
  - 1235.6.44006 Boehringer Ingelheim Investigational Site, Whitstable

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Started | 315 | 315 | 317
Completed | 301 | 297 | 307
Not Completed | 14 | 18 | 10
Not completed — Adverse Event | 8 | 10 | 5
Not completed — Non compliant with protocol | 3 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Consent withdrawn | 2 | 3 | 1
Not completed — Specified category | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg | Total
Number analyzed (Participants) | 315 | 315 | 317 | 947
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (10.4) | 57.6 (9.4) | 55.5 (9.8) | 56.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 145 | 146 | 419
  Male | 187 | 170 | 171 | 528

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure
Description: Change from baseline to the end of study in trough DBP
Time Frame: Baseline and end of study (8 weeks or last value on treatment)
Population: Full analysis set of patients who had a baseline trough blood pressure measurement and at least one post baseline trough blood pressure measurement using last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
mmHg | -6.48 (0.45) | -9.24 (0.45) | -9.33 (0.45)
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Testing that the combination treatments are superior to monotherapy A10. The number of patients in the treatment arms ensure the tests have over 90% power; Test type: Superiority or Other; p < 0.0001, ANCOVA — Doses tested against A10 in a hierarchical manner to address issues of multiplicity. T80/A10 was tested first, then T40/A10; Adjusted for baseline and country effect; Least Squares Mean Difference = -2.76, 95% CI [-3.77 to -1.75], Standard Error of Mean 0.52
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted for baseline and country effect; Least Squares Mean Difference = -2.85, 95% CI [-3.86 to -1.84], Standard Error of Mean 0.51

2. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure
Description: Change from baseline to the end of study in trough SBP
Time Frame: Baseline and end of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
mmHg | -7.44 (0.66) | -11.09 (0.66) | -11.29 (0.66)
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -3.66, 95% CI [-5.15 to -2.16], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -3.85, 95% CI [-5.35 to -2.36], Standard Error of Mean 0.76

3. Secondary Outcome: Trough Seated Diastolic Blood Pressure Control (Defined as < 90mmHg)
Description: The number of patients who reach the target DBP of <90mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Yes (DBP<90 mmHg) | 156 | 195 | 206
  No (DBP>=90 mmHg) | 149 | 111 | 104
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.002, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.21 to 2.32]
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.91, 95% CI [1.37 to 2.65]

4. Secondary Outcome: Trough Seated Diastolic Blood Pressure <80 mmHg
Description: The number of patients who reach the target DBP of <80mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Yes (DBP<80 mmHg) | 18 | 39 | 39
  No (DBP>=80 mmHg) | 287 | 267 | 271
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.004, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 2.35, 95% CI [1.30 to 4.25]
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.004, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 2.33, 95% CI [1.29 to 4.22]

5. Secondary Outcome: Trough Seated DBP Response
Description: The number of patients who reach the target DBP of <90mmHg or had a reduction in DBP >= 10mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Yes (Responder) | 163 | 202 | 213
  No (Non-responder) | 142 | 104 | 97
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.002, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.68, 95% CI [1.21 to 2.34]
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.92, 95% CI [1.38 to 2.68]

6. Secondary Outcome: Trough Seated SBP Control
Description: The number of patients who reach the target SBP of <140mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Yes (SBP<140 mmHg) | 153 | 180 | 187
  No (SBP>=140 mmHg) | 152 | 126 | 123
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.027, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.44, 95% CI [1.04 to 2.00]
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.008, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.55, 95% CI [1.12 to 2.15]

7. Secondary Outcome: Trough Seated SBP Response
Description: The number of patients who reach the target SBP of <140mmHg or had a reduction in SBP >= 15 mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Yes (Responder) | 165 | 198 | 204
  No (Non-responder) | 140 | 108 | 106
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.006, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.58, 95% CI [1.14 to 2.21]
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.002, Mantel Haenszel; Mantel-Haenszel statistics adjusted for country effect; Odds Ratio (OR) = 1.67, 95% CI [1.20 to 2.32]

8. Secondary Outcome: Trough Seated BP Normality Classes
Description: The number of patients who reach predefined BP categories
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Participants
  Optimal (SBP<120 and DBP<80 mmHg) | 0 | 12 | 6
  Normal (SBP<130 and DBP<85 mmHg and not optimal) | 36 | 43 | 50
  High-normal (SBP<140 DBP<90 mmHg and not normal) | 77 | 91 | 106
  Stage 1 hypertension (SBP<160 and DBP<100 mmHg) | 157 | 139 | 133
  Stage 2 hypertension (SBP>=160 and DBP>=100 mmHg) | 35 | 21 | 15
Statistical Analysis 1: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 10mg; Test type: Superiority or Other; p = 0.006, Wilcoxon rank sum test; Stratified (for country) Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 10mg; Test type: Superiority or Other; p < 0.001, Wilcoxon rank sum test; Stratified (for country) Wilcoxon rank sum test

9. Secondary Outcome: Oedema Incidence Rate
Description: The number of patients who experienced at least one case of oedema or worsening of oedema for the first time (expressed as number of patients/100 patient-years)
Time Frame: During randomised treatment period
Population: as for outcome 1
Measure: Number; unit: Number of patients/100 patient-years
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Number of patients/100 patient-years | 44.7 | 42.8 | 54.0

10. Secondary Outcome: Peripheral Oedema Incidence Rate
Description: The number of cases of peripheral oedema (expressed as number of cases/100 patient-years)
Time Frame: During randomised treatment period
Measure: Number; unit: Number of cases/100 patient-years
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Number analyzed (Participants) | 305 | 306 | 310
Number of cases/100 patient-years | 48.8 | 44.8 | 54.0

ADVERSE EVENTS:
Arm/Group | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Serious Adverse Events (participants affected / at risk) | 1 | 3 | 0
Other Adverse Events (participants affected / at risk) | 22 | 21 | 27
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Cardiac failure (Cardiac disorders) | 0/315 | 1/315 | 0/317
Local swelling (General disorders) | 0/315 | 1/315 | 0/317
Bronchitis (Infections and infestations) | 1/315 | 0/315 | 0/317
Ruptured cerebral aneurysm (Nervous system disorders) | 0/315 | 1/315 | 0/317
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 10mg | Telmisartan 80mg and Amlodipine 10mg
Peripheral oedema (General disorders) | 22/315 | 21/315 | 27/317

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.